CLINICAL TRIAL: NCT04509999
Title: Randomized Trial of Bicalutamide to Block TMPRSS2 in Males With COVID-19 Infection
Brief Title: Bicalutamide to Block TMPRSS2 in Males With COVID-19 Infection
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No patients enrolled and funding withdrawn
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB202001669-A; OCR38162 (Other: UF OnCore)
Record Dates: First submitted 2020-08-07; First posted 2020-08-12 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — bicalutamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of care and Experimental treatment of Bicalutamide (Experimental): Each subject will be administered bicalutamide 150 mg daily at 1:1 randomization for up to 4 weeks.
  Interventions: Drug: Bicalutamide 150 Mg Oral Tablet
- Standard of Care and Placebo (Placebo Comparator): Each subject will be administered placebo as formulated at 1:1 randomization for up to 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bicalutamide 150 Mg Oral Tablet — Bicalutamide 150 mg by mouth daily
  Arms: Standard of care and Experimental treatment of Bicalutamide
Drug: Placebo — Placebo as formulated by mouth daily
  Arms: Standard of Care and Placebo

SUMMARY:
COVID-19 outcomes are worse in male patients. Androgen signaling, therefore, is a target for clinical exploration. TMPRSS2 is a membrane protease required for COVID pathogenesis that is regulated by androgens. Blocking TMPRSS2 with bicalutamide may reduce viral replication and improve the clinical outcome. Therefore, the study proposes to test bicalutamide at 150 mg oral daily dosing in a double-blind placebo-controlled randomized trial in male patients with early symptomatic COVID-19 disease.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be eligible for study participation:

* Men ≥ 36 years old diagnosed with at least one temperature elevation ≥ 100.4 F., OR new cough, OR new dyspnea AND documented COVID-19 positive by approved standard local laboratory assay
* Men ≥ 18 years but < 36 years old must exhibit EITHER new cough, OR new dyspnea AND documented COVID-19 positive by approved standard local laboratory assay.
* Access to working telephone or other form of communication such as email.
* Randomization within 7 days of COVID-positive study result. All subjects will undergo repeat COVID-19 assay on day 0 enrollment and a positive test is required to stay on study
* Written informed consent obtained from the subject and the subject agrees to comply with all study-related procedures

Exclusion Criteria:

Subjects with any of the following will not be eligible for study participation:

* Randomization greater than 7 days from a positive COVID test result. All subjects will undergo repeat COVID-19 assay on day 0 enrollment and a negative test will result in a screen-fail and removal from study
* Admission to hospital at time of screening
* Inclusion in another randomized trial for COVID therapy
* Diagnosis of prostate cancer and/or treatment with anti-androgen in the past 3 months
* Current treatment with any androgen replacement products
* Prior allergic reaction or intolerance to Bicalutamide or other Androgen receptor Inhibitors
* Requirement for coumarin product or warfarin products due to potential displacement by bicalutamide
* Subject unable to take oral bicalutamide
* Known Hepatitis B or C
* Liver Cirrhosis
* AST/ALT greater than or equal to 3 X institutional ULN

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only men > 18 years of age are eligible for this trial testing anti-androgen agents. This medication has not been approved for use in women.
Enrollment: 0 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion x 100 = percent of patients with improved COVID-19 symptoms | Day 28
  COVID-19 symptom relief at day 28, and % of COVID-19 symptom relief and its 95% confidence interval (CI) will be calculated using the exact binomial distribution and compared using Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Kaye, MD, Principal Investigator — University of Florida

IPD SHARING:
Plan to Share IPD: No